CLINICAL TRIAL: NCT02221570
Title: A Randomized Placebo Controlled Study of Baclofen in the Treatment of Muscle Cramps in Patients With Cirrhosis
Brief Title: Baclofen in the Treatment of Muscle Cramps in Patients With Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ibrahim Shebl, Dr., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: baclofen cramps
Record Dates: First submitted 2014-08-14; First posted 2014-08-20 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Muscle Cramps; Liver Cirrhosis
MeSH Terms: conditions — Muscle Cramp; Liver Cirrhosis | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Baclofen (Active Comparator): Baclofen, a derivative of gamma-aminobutyric acid, is a muscle relaxant and an antispastic agent. It was introduced in 1966 as a possible treatment for spasticity due to corticospinal tract lesions. Baclofen was also tested with promising results in the treatment of other medical disorders such as cluster headaches, gastroesophageal reflux disease,chronic hiccups and cough.
  Interventions: Drug: Baclofen
- Placebo (Placebo Comparator): placebo of baclofen

INTERVENTIONS:
Drug: Baclofen — Baclofen, a derivative of gamma-aminobutyric acid, is a muscle relaxant and an antispastic agent. It was introduced in 1966 as a possible treatment for spasticity due to corticospinal tract lesions. Baclofen was also tested with promising results in the treatment of other medical disorders such as cluster headaches, gastroesophageal reflux disease,chronic hiccups and cough.
  Other Names: Gablofen; Lioresal; Apo-Baclofen; Dom-Baclofen; Liotec; Med-Baclofen; Mylan-Baclofen; Novo-Baclofen; Nu-Baclo; PHL-Baclofen; PMS-Baclofen; ratio-Baclofen; Riva-Baclofen
  Arms: Baclofen

SUMMARY:
Patients with cirrhosis often experience muscle cramps with varying severity. The mechanism of their occurrence is not yet understood. Muscle cramps in patients with cirrhosis are associated with significantly diminished quality of life.

The aim of the study is to assess the efficacy of baclofen in the treatment of muscle cramps in patients with liver cirrhosis.

DETAILED DESCRIPTION:
Muscle cramps are common in patients with liver disease and associated with significantly diminished quality of life. Patients with cirrhosis often experience muscle cramps with varied frequency and severity. The exact mechanisms by which they occur remain unclear, although a number of pathophysiological events unique to liver disease may contribute. Clinical studies have identified alterations in 3 areas: nerve function, energy metabolism, and plasma volume/electrolytes.

Although a number of mechanisms for cramps in liver disease have been postulated and have been targeted by medical therapies, a clear picture of the causal events has not emerged. Several agents as vitamin E, human albumin, zinc, taurine, eperisone hydrochloride and branched-chain amino acids have shown some benefit in small uncontrolled studies, although large randomized controlled trials are lacking.

Baclofen, a derivative of gamma-aminobutyric acid, is a muscle relaxant and an antispastic agent. It was introduced in 1966 as a possible treatment for spasticity due to corticospinal tract lesions. Baclofen was also tested with promising results in the treatment of other medical disorders such as cluster headaches, gastroesophageal reflux disease,chronic hiccups and cough.

The aim of the study is to assess the efficacy of baclofen in the treatment of muscle cramps in patients with liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis
* Muscle cramps( ≥3 cramps per week )

Exclusion Criteria:

* Allergy to baclofen
* Renal impairment
* Pregnant and lactating women
* Peripheral vascular disease
* Peripheral neuropathy
* Medications as calcium channel blockers, conjugated estrogens and naproxen.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with decreased incidence of muscle cramps after taking Baclofen compared with placebo. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Asem A Elfert, MD, Principal Investigator — Tanta Faculty of Medicine, Professor; Lobna A AboAli, Study Director — Tanta Faculty of Medicine, Lecturer; Samah M Soliman, Study Director — Tanta Faculty of Medicine, Lecturer; Ibrahim Shebl, Study Director — Tanta University Hospitals, House Officer
Locations (1):
- Tanta University Hospital, Tanta, Gharbia Governorate, Egypt

REFERENCES:
- [Background] Chatrath H, Liangpunsakul S, Ghabril M, Otte J, Chalasani N, Vuppalanchi R. Prevalence and morbidity associated with muscle cramps in patients with cirrhosis. Am J Med. 2012 Oct;125(10):1019-25. doi: 10.1016/j.amjmed.2012.03.012. Epub 2012 Jul 24. PMID 22835465
- [Background] Mehta SS, Fallon MB. Muscle cramps in liver disease. Clin Gastroenterol Hepatol. 2013 Nov;11(11):1385-91; quiz e80. doi: 10.1016/j.cgh.2013.03.017. Epub 2013 Mar 28. PMID 23542334
- [Background] Hudgson P, Weightman D. Baclofen in the treatment of spasticity. Br Med J. 1971 Oct 2;4(5778):15-7. doi: 10.1136/bmj.4.5778.15. PMID 4938243
- [Background] Hering-Hanit R, Gadoth N. The use of baclofen in cluster headache. Curr Pain Headache Rep. 2001 Feb;5(1):79-82. doi: 10.1007/s11916-001-0014-1. PMID 11252142
- [Background] Orr WC, Goodrich S, Wright S, Shepherd K, Mellow M. The effect of baclofen on nocturnal gastroesophageal reflux and measures of sleep quality: a randomized, cross-over trial. Neurogastroenterol Motil. 2012 Jun;24(6):553-9, e253. doi: 10.1111/j.1365-2982.2012.01900.x. Epub 2012 Mar 8. PMID 22404184
- [Background] Burke AM, White AB, Brill N. Baclofen for intractable hiccups. N Engl J Med. 1988 Nov 17;319(20):1354. doi: 10.1056/NEJM198811173192016. No abstract available. PMID 3185643
- [Background] Froestl W. Chemistry and pharmacology of GABAB receptor ligands. Adv Pharmacol. 2010;58:19-62. doi: 10.1016/S1054-3589(10)58002-5. PMID 20655477